CLINICAL TRIAL: NCT05183438
Title: Construction of a Prediction Model for Metachronous Colorectal Adenoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-SR-343
Record Dates: First submitted 2021-12-26; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Metachronous Colorectal Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with metachronous colorectal adenomas
- patients without metachronous colorectal adenomas

SUMMARY:
The study aimed to explore the independent risk factors for the metachronous colorectal adenoma after endoscopic resection, and construct the prediction model of metachronous colorectal adenoma, in order to provide theoretical basis for postoperative follow-up time of patients, and allocate limited medical resources.

DETAILED DESCRIPTION:
A large cohort of eligible patients were included in the analysis, and classified into derivation and validation cohorts at a ratio of 7:3. Demographic and clinicopathological characteristics of participants were utilized to develop a prediction model for metachronous colorectal adenoma. In the derivation cohort, the LASSO regression method was applied to filter variables and multivariate logistic regression analysis was used to identify important predictors.A prediction model was established based on the results of multivariate logistic regression analysis. The predictive performance of the model was evaluated with respect to its discrimination, calibration and clinical usefulness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 and ≤75 years old. Patients with complete data on demography and clinicopathology.

Exclusion Criteria:

* Patients with a history of inflammatory bowel disease, enterophthisis, familial adenomatous polyposis, P-J syndrome and intestinal lymphoma.

Patients with a previous history of colorectal neoplasm. Patients with a history of severe systemic diseases. Lack of complete clinical data for analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed eligible patients, 18 to 75 years of age, including cases with metachronous colorectal adenomas and controls without metachronous colorectal adenomas, are enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics of patients with metachronous colorectal adenomas checklist | 3 year
  Age (years), sex (man/woman), family history of colorectal cancer (in first-degree relatives, including parents and siblings), history of smoking (never, past, current), history of alcohol consumption (never, past, current), regular use of non-steroidal anti-inflammatory drugs

SECONDARY OUTCOMES:
Cumulative recurrence rate of metachronous colorectal adenomas | 3 year
  Cumulative recurrence rate

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta S, Lieberman D, Anderson JC, Burke CA, Dominitz JA, Kaltenbach T, Robertson DJ, Shaukat A, Syngal S, Rex DK. Recommendations for Follow-Up After Colonoscopy and Polypectomy: A Consensus Update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1131-1153.e5. doi: 10.1053/j.gastro.2019.10.026. Epub 2020 Feb 7. No abstract available. PMID 32044092